CLINICAL TRIAL: NCT05108857
Title: PET Imaging of Systemic Sclerosis Using 18F-FDG and 68Ga-DOTA-Siglec-9
Brief Title: PET Imaging of Systemic Sclerosis Using FDG and 68Ga-DOTA-Siglec-9
Acronym: SYSPET
Status: Enrolling by invitation | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Collaborators: Kuopio University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2110/2021
Record Dates: First submitted 2021-10-25; First posted 2021-11-05 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Skin biopsies Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study evaluates the potential of positron emission tomography (PET)/computed tomography (CT) imaging to monitor disease activity in patients with systemic sclerosis (SSc). PET/CT imaging will focus on two pathological features of SSc, i.e. metabolic activity evaluated by glucose analog 18F-FDG, and expression of inflammation-inducible vascular adhesion protein 1 (VAP-1) evaluated by 68Ga-DOTA-Siglec-9 tracer.

DETAILED DESCRIPTION:
In patients with systemic sclerosis (SSc), the quantitative assessment of disease activity is still difficult. Identification of patients who unlikely respond to therapy before or early in a course of the treatment could reduce morbidity and produce cost-savings. This project will evaluate the potential of advanced functional imaging techniques to monitor disease activity. Functional imaging will focus on two pathological features of SSc, i.e. metabolic activity evaluated by glucose analog 18F-FDG positron emission tomography (PET)/computed tomography (CT), and expression of inflammation-inducible vascular adhesion protein 1 (VAP-1) evaluated by new 68Ga-DOTA-Siglec-9 tracer. If successful, the resulting techniques may prove invaluable as tools in the clinical practice and in drug research aiming to find new targets to the treatment of SSc.

ELIGIBILITY:
Inclusion Criteria:

* Adults with active systemic sclerosis (SSc).
* Onset of SSc (defined as first non-Raynaud symptom) not more than 5 years ago.
* Clinically active disease with proximal nailfold capillary abnormalities detected with videocapillaroscopy and/or raised inflammatory markers (CRP or ESR).

Exclusion Criteria:

* Underage, pregnant, breastfeeding, handicapped or prisoner
* History of or current inflammatory joint disease or autoimmune disease other than SSc.
* History of treatment with, prior to this study, immunosuppressives or disease-modifying anti-rheumatic drugs (DMARDs) such as methotrexate, leflunomide, azathioprine, mycophenolate, cyclophosphamide or biologic agents such as anti-TNF inhibitors, abatacept, or rituximab. Hydroxychloroquine is allowed in the history (≥3 months prior to PET study).
* Intra-articular or parenteral corticosteroids ≤4 weeks prior to PET/CT study.
* Prostanoids or other vasoactive treatments like phosphodiesterase-5 inhibitors or endothelin receptor antagonists ≤4 weeks prior to PET/CT study (the use of calcium channel inhibitors is allowed).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of Turku University Hospital or Kuopio University Hospital with active systemic sclerosis.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2021-11-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection of inflammation in PET/CT images | Day 1
  Standardized uptake value of PET tracer at the sites of inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Anne Roivainen, Principal Investigator — Turku University Hospital, Turku PET Centre
Locations (1):
- Turku University Hospital, Turku PET Centre, Turku, Finland